CLINICAL TRIAL: NCT01506284
Title: Assessment of Airways Mechanical Properties by Forced Oscillatory Technique (FOT) and Laser Interferometry (LIR) During Anesthesia.
Brief Title: Assessment of Airways Mechanical Properties by FOT and LIR During Anesthesia
Status: Completed | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Peter Kostic, Principal investigator, Uppsala University Hospital
Other Study IDs: Uppsala 2011 - 189
Record Dates: First submitted 2011-12-09; First posted 2012-01-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2012-01

CONDITIONS: Anesthesia
Keywords: Forced oscillatory technique; Laser interferometry; Intravenous anesthesia; Mechanical ventilation; Pressure controlled ventilation; Airways mechanical properties; Respiratory system reactance; Oscillatory mechanics; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anesthetized patients ASA I-II: ASA classification I-II, scheduled for elective surgery requiring general anesthesia.
  Interventions: Procedure: Forced oscillatory technique (FOT) and laser interferometry (LIR).

INTERVENTIONS:
Procedure: Forced oscillatory technique (FOT) and laser interferometry (LIR). — FOT: The stimulating signal is generated by an A/D-D/A board and amplified by a power amplifier that drives a loudspeaker the output of which is connected to inspiratory line of the ventilator. Pressure and flow are measured at the inlet of the endotracheal tube by a piezoresistive pressure transducer and a mesh-type heated pneumotachograph coupled with a differential pressure transducer.
  LIR: The scanner unit is made by three laser interferometers, the beams of which are deflected on the chest wall surface by a mirror moved by a stepper motor triggered on the respiratory pattern of patient.

SUMMARY:
The aims of the present study are:

1. To evaluate the effect of the induction of anaesthesia and paralysis in terms of changes in oscillatory mechanics parameters
2. To evaluate the mechanical properties of the respiratory system in terms of input and transfer oscillatory impedance in response to PEEP changes

DETAILED DESCRIPTION:
It has been recently shown that respiratory system reactance (Xrs) obtained by the forced oscillation technique (FOT) at 5 Hz is more reliable than dynamic compliance for assessing lung collapse and the effects of lung RMs in a porcine ALI model ( Ref.1,2).

Specifically, Xrs (and its derived variable CX5, the oscillatory compliance at 5 Hz) identifies the minimum positive end-expiratory pressure (PEEP) level required to maintain lung recruitment with high sensitivity and specificity. Moreover, it has been recently demonstrated that Xrs may be used to identify the lowest level of PEEP able to prevent atelectasis and that PEEP setting strategy based on maximizing Xrs is able to limit lung injury compared to oxygenation-based approach in a porcine lavage model of lung injury. ( Ref.3)

Recently, at the biomedical engineering department of Politecnico di Milano measurements of chest wall displacement have been successfully performed by means of an optical sensor realized using a laser self-mixing interferometer (LIR). The advantage of this approach is that it is contact-less, that by deflecting the laser been it is possible to scan any region of the chest wall surface and that it allows to measure also low-frequency vibrations.

Protocol

1. The baseline pulmonary function will be assessed by spirometry before surgery.
2. Just before surgery measurements of oscillatory mechanics will be performed at the following stages:

   * awake patient
   * spontaneous ventilation through the laryngeal mask after induction of anesthesia
   * pressure controlled ventilation (PCV) after the administration of neuromuscular blocking agent and intubation and PEEP 0 cmH2O
   * PCV with PEEP 5 cmH2O
   * Recruitment maneuver (RM) (peak pressure 30 cmH2O and PEEP 15 cmH2O) for 2 minutes
   * PCV with PEEP 5 cmH2O after RM

At each stage the following measurements will be performed:

* Input impedance at 5-11-19 Hz by FOT
* the movements of the chest wall assessed by laser interferometry (LIR) applying two different stimulating waveforms: 5-11-19 Hz and 100 Hz
* functional residual capacity (FRC)
* arterial blood gas measurement (ABG)

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* ASA I-II, scheduled for elective surgery requiring general anesthesia
* signed informed consent

Exclusion Criteria:

* patient refusal
* BMI > 35
* co-existing respiratory disease (COPD, asthma, restrictive lung disease)
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ASA classification I-II, scheduled for elective surgery requiring general anesthesia
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in respiratory system impedance | baseline and 5 minutes of ventilation
  FOT measurements:
  Respiratory system impedance will be computed from the flow and pressure signals measured at the inlet of the tracheal tube. A composite waveform including 5, 11 and 19 Hz will be used as a stimulating signal generated by an A/D-D/A board and amplified by a power amplifier that drives a loudspeaker the output of which is connected to inspiratory line of the ventilator.

SECONDARY OUTCOMES:
Change in chest wall displacement measured by LIR | baseline and 5 minutes of ventilation
  Laser interferometry (LIR):
  The movement of 18 points of the chest wall will be measured by a self-mixing interferometer. The measurement points will be chosen along three vertical lines (the midline and the two parasternal lines) and will be equally distributed from the clavicles to the anterior superior iliac spines. The chest wall movement will be measured in response to two different stimulating waveforms: a composite waveform including 5, 11 and 19 Hz, a sinusoidal signal at 100 Hz.
Change in oxygenation (paO2) | baseline and 5 minutes of ventilation
  Arterial blood gas measurement (ABG)
Change in Functional residual capacity (FRC) | baseline and 5 minutes of ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Frykholm, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hopsital, Dep. of Anesthesia and Intensive Care, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Background] Dellaca RL, Andersson Olerud M, Zannin E, Kostic P, Pompilio PP, Hedenstierna G, Pedotti A, Frykholm P. Lung recruitment assessed by total respiratory system input reactance. Intensive Care Med. 2009 Dec;35(12):2164-72. doi: 10.1007/s00134-009-1673-3. Epub 2009 Sep 30. PMID 19789855
- [Background] Dellaca RL, Zannin E, Kostic P, Olerud MA, Pompilio PP, Hedenstierna G, Pedotti A, Frykholm P. Optimisation of positive end-expiratory pressure by forced oscillation technique in a lavage model of acute lung injury. Intensive Care Med. 2011 Jun;37(6):1021-30. doi: 10.1007/s00134-011-2211-7. Epub 2011 Apr 1. PMID 21455750
- [Background] Kostic P, Zannin E, Andersson Olerud M, Pompilio PP, Hedenstierna G, Pedotti A, Larsson A, Frykholm P, Dellaca RL. Positive end-expiratory pressure optimization with forced oscillation technique reduces ventilator induced lung injury: a controlled experimental study in pigs with saline lavage lung injury. Crit Care. 2011;15(3):R126. doi: 10.1186/cc10236. Epub 2011 Apr 28. PMID 21575220